CLINICAL TRIAL: NCT01398319
Title: Prevention of Alcohol Related Incidents in the US Air Force
Acronym: AFIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH); United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melissa Little, PhD, MPH, Associate Professor, Department of Public Health Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FWH20140105H
Record Dates: First submitted 2011-07-11; First posted 2011-07-20 (Estimated); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Abuse
Keywords: prevention; alcohol abuse
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Brief Alcohol Booster Intervention (Experimental): The 1-hour booster intervention was delivered using MI to extend the effective elements found in the original BAI intervention with elements from behavioral economic theory. A behavioral economic approach to alcohol use suggests that decisions to drink are more likely when 1) there is a lack of access to or engagement in alternative alcohol-free reinforcing activities, and 2) there is a greater relative focus on immediate, relative to delayed, rewards (i.e., steep delayed reward discounting). The intent of the intervention is to bring important long-term goals into the present so that the immediate awareness of this goal might diminish the relative benefit of drinking. Another goal was to have the Airmen identify enjoyable and goal-consistent alcohol-free activities they could engage in during their free time. The booster also included a reminder of the U.S. Air Forces rules and policies on alcohol use and harm reduction drinking strategies.
  Interventions: Behavioral: Group Brief Alcohol Intervention; Behavioral: Group Brief Alcohol Intervention Booster
- Bystander Intervention (Active Comparator): The 1-hour Bystander intervention was a non-alcohol related briefing that served as the control condition. The intervention focused on increasing Airmen's awareness of the qualities of being a good "wingman" (e.g., watching for their peers) and how those are tied to the Air Force Core Values. It aimed to increase participants' perceived responsibility to act in certain situations. The intervention draws on the philosophy that members in a community have a role in shifting social norms to prevent violence. While the intervention did not directly discuss alcohol use, the focus on military values and taking responsibility for one's self and others could contribute to healthier drinking-related choices.
  Interventions: Behavioral: Group Brief Alcohol Intervention; Behavioral: Bystander Intervention

INTERVENTIONS:
Behavioral: Group Brief Alcohol Intervention — The BAI contained components of effective interventions developed for young adult drinkers both in health care and educational settings and was specifically tailored to the unique needs and risk factors of Airmen. The 1-hour group intervention was administered using the principles of motivational interviewing (MI) in an interactive Socratic style to generate feedback and discussion. Open-ended questions, reflections, as well as the decisional balance scale were used to increase Airmen's motivation to remain alcohol free.
Behavioral: Group Brief Alcohol Intervention Booster — The 1-hour booster intervention was delivered using MI to extend the effective elements found in the original BAI intervention with elements from behavioral economic theory. A behavioral economic approach to alcohol use suggests that decisions to drink are more likely when 1) there is a lack of access to or engagement in alternative alcohol-free reinforcing activities, and 2) there is a greater relative focus on immediate, relative to delayed, rewards (i.e., steep delayed reward discounting). The intent of the intervention is to bring important long-term goals into the present so that the immediate awareness of this goal might diminish the relative benefit of drinking. Another goal was to have the Airmen identify enjoyable and goal-consistent alcohol-free activities they could engage in during their free time. The booster also included a reminder of the U.S. Air Forces rules and policies on alcohol use and harm reduction drinking strategies.
  Other Names: Making Responsible Choices
  Arms: Group Brief Alcohol Booster Intervention
Behavioral: Bystander Intervention — The 1-hour Bystander intervention was a non-alcohol related briefing that served as the control condition. The intervention focused on increasing Airmen's awareness of the qualities of being a good "wingman" (e.g., watching for their peers) and how those are tied to the Air Force Core Values. It aimed to increase participants' perceived responsibility to act in certain situations. The intervention draws on the philosophy that members in a community have a role in shifting social norms to prevent violence (Coker et al., 2011). While the intervention did not directly discuss alcohol use, the focus on military values and taking responsibility for one's self and others could contribute to healthier drinking-related choices.
  Arms: Bystander Intervention

SUMMARY:
Alcohol misuse poses significant public health concerns in the U.S. military. A Brief Alcohol Intervention (BAI) have been shown to reduce alcohol related incidents among Airmen undergoing training. The current study sought to examine whether a booster BAI administered at the end of an Airmen's training reduced alcohol related incidents out to a one-year follow-up. Participants were 26,231 US Air Force Technical Trainees recruited between March 2016 and July 2018. Participants were cluster randomized by cohort to two conditions: BAI + BAI Booster or BAI + Bystander Intervention. The primary analysis was a comparison of the interventions' efficacies in preventing Article 15 alcohol related incidents at a one-year follow-up, conducted using a generalized estimating equations logistic regression model controlling for covariates.

ELIGIBILITY:
Participants were Airmen undergoing Technical Training at five military bases (Lackland Air Force Base, Keesler Air Force Base, Sheppard Air Force Base, Goodfellow Air Force Base and Fort Sam Houston) in Texas and Mississippi from March 2016 through July 2018. Eligibility criteria included being at least 18 years of age and understanding the consent process in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26231 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Article 15s | 12 months
  Adjudicated alcohol related incident in the United States Air Force (Article 15). We determined if an Airmen had received an Article 15 in the year following Technical Training by searching the Automated Military Justice Analysis and Management System (AMJAMS).

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Klesges, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- 37th Training Group, Lackland Air Force Base, Texas, United States